CLINICAL TRIAL: NCT05556343
Title: A Phase 2a, Open-label, Pilot Study to Evaluate Efficacy, Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of MYK-224 in Participants With Symptomatic Hypertrophic Cardiomyopathy and Left Ventricular Outflow Tract Obstruction (MERCUTIO)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of MYK-224 in Participants With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Acronym: MERCUTIO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV029-009; 2022-001292-14 (EudraCT Number); U1111-1276-3555 (Registry Identifier: WHO)
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: Obstructive Hypertrophic Cardiomyopathy; MYK-224; BMS-986435; HCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive MYK-224 either as a monotherapy or in combination with standard-of-care consisting of a beta-blocker. Participants who complete Cohort 1 will be eligible for an optional open label extension period
  Interventions: Drug: MYK-224
- Cohort 2 (Experimental): Participants will receive MYK-224 in combination with standard-of-care consisting of either a calcium channel blocker or disopyramide (which is given in combination with either a beta-blocker or calcium channel blocker). Participants who complete Cohort 2 will be eligible for an optional open label extension period
  Interventions: Drug: MYK-224

INTERVENTIONS:
Drug: MYK-224 — Specified dose on specified days
  Other Names: BMS-986435

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of MYK-224 in participants with obstructive Hypertrophic Cardiomyopathy (oHCM)

ELIGIBILITY:
Inclusion Criteria:

* Has adequate acoustic windows, to enable accurate TTEs as determined by the echocardiography core laboratory.
* Men or women diagnosed with oHCM consistent with current American College of Cardiology Foundation/American Heart Association and European Society of Cardiology guidelines, satisfying both of the following criteria:

  * Has unexplained left ventricular (LV) hypertrophy with nondilated ventricular chambers in the absence of other cardiac (eg, hypertension, aortic stenosis) or systemic disease and with maximal LV wall thickness ≥ 15 millimeter (mm) (or ≥ 13 mm with positive family history of hypertrophic cardiomyopathy or with a known disease-causing mutation), as determined by core laboratory interpretation.

AND

-- Has a LVOT peak gradient during screening as assessed by echocardiography of ≥ 50 millimeters of mercury (mm Hg) at rest, or ≥ 30 mm Hg at rest and ≥ 50 mm Hg with Valsalva maneuver (confirmed by echocardiography core laboratory interpretation).

* Has resting LVEF ≥ 60% at the Screening visit as determined by echocardiography core laboratory.
* New York Heart Association (NYHA) functional class II or III symptoms at screening.
* Has a valid measurement of LVOT post-exercise peak gradient at screening as determined by echocardiography core laboratory.

Exclusion Criteria:

* Presence of any medical condition that precludes exercise stress testing.
* History of syncope or sustained ventricular tachyarrhythmia within 6 months prior to screening.
* Known infiltrative or storage disorder causing cardiac hypertrophy that mimics HCM, such as Fabry disease, amyloidosis, or Noonan syndrome with left ventricular hypertrophy.
* Prior treatment with mavacamten or aficamten. An exception may be made in cases where myosin inhibitor use was not within 4 months of the Screening visit, and with the agreement of both the Investigator and the Medical Monitor.
* Has been successfully treated with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA]) within 6 months prior to Screening or plans to have either of these treatments during the study (Note: Individuals with an unsuccessful myectomy or percutaneous ASA procedure performed > 6 months prior to Screening may be enrolled if study eligibility criteria for LVOT gradient criteria are met).
* Implantable cardioverter-defibrillator (ICD) placement or pulse generator change within 2 months prior to screening or planned new ICD placement during the study (pulse generator changes, if needed during the study are allowed).
* Has a history of resuscitated sudden cardiac arrest (any time) or known history of appropriate implantable cardioverter-defibrillator (ICD discharge for life-threatening ventricular arrhythmia within 6 months prior to screening.
* Has paroxysmal, atrial fibrillation with atrial fibrillation present per the Investigator's evaluation of the participant's ECG at the time of Screening.
* Has persistent or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to Screening and/or not adequately rate controlled within 6 months prior to Screening (Note: Participants with persistent or permanent atrial fibrillation who are anticoagulated and adequately rate-controlled are allowed).
* Has QT interval with Fridericia correction (QTcF) > 500 msec when QRS interval < 120 msec or QTcF > 520 msec when QRS ≥ 120 msec if participant has left bundle branch block or any other 12-lead ECG abnormality considered by the investigator to pose a risk to participant safety (eg, second-degree atrioventricular block type II).
* Has known moderate or severe (per investigator's judgment) aortic valve stenosis at screening.
* History of LV systolic dysfunction (LVEF < 45%) at any time during their clinical course.
* Clinically significant pulmonary disease associated with exertional dyspnea.
* Has known significant unrevascularized obstructive coronary artery disease (>70% stenosis in one or more main epicardial coronary arteries) or history of myocardial infarction Note: participants with prior coronary artery bypass grafting (CABG) or percutaneous coronary interventions (PCIs) are allowed if the procedure was performed at least 12 weeks prior to screening
* Prior treatment with cardiotoxic agents such as anthracyclines (eg, doxorubicin) or similar

Other protocol-defined criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 53 weeks
Incidence of arrhythmias | Up to 53 weeks
Incidence of appropriate implantable cardioverter defibrillator therapy and resuscitated cardiac arrest | Up to 53 weeks
Incidence of vital sign abnormalities | Up to 53 weeks
Incidence of physical examination abnormalities | Up to 53 weeks
Incidence of electrocardiogram (ECG) abnormalities | Up to 53 weeks
Incidence of transthoracic echocardiogram (TTE) abnormalities | Up to 53 weeks
Incidence of clinical laboratory abnormalities | Up to 53 weeks

SECONDARY OUTCOMES:
Change in left ventricular outflow tract (LVOT) peak gradient (post-exercise, resting, and Valsalva) from baseline to end of treatment | Up to 45 weeks
Proportion of participants achieving a resting LVOT peak gradient of < 30 mm Hg and a Valsalva LVOT peak gradient < 50 mm Hg at end of treatment | Up to 45 weeks
Concentration-response relationship between MYK-224 pharmacokinetics (PK) and LVOT peak gradients | Up to 45 weeks
Concentration-response relationship between MYK-224 PK and echocardiographic parameters of systolic and diastolic function | Up to 45 weeks
Summary of plasma concentrations of MYK-224 | Up to 53 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- United States (12):
  - Local Institution - 0026, La Jolla, California
  - Local Institution - 0014, Los Angeles, California
  - Local Institution - 0016, San Francisco, California
  - Local Institution - 0001, Kansas City, Kansas
  - Local Institution - 0032, New York, New York
  - Local Institution - 0013, Durham, North Carolina
  - Local Institution - 0031, Cincinnati, Ohio
  - Local Institution - 0015, Cleveland, Ohio
  - Local Institution - 0024, Portland, Oregon
  - Local Institution - 0021, Nashville, Tennessee
  - Local Institution - 0025, San Antonio, Texas
  - Local Institution - 0006, Salt Lake City, Utah
- Italy (3):
  - Local Institution - 0027, Bologna, BO
  - Local Institution - 0005, Florence, FI
  - Local Institution - 0029, Milan
- Poland (2):
  - Local Institution - 0011, Katowice, Silesian Voivodeship
  - Local Institution - 0030, Wroclaw
- Spain (8):
  - Local Institution - 0028, Alicante, A
  - Local Institution - 0022, Granada, GR
  - Local Institution - 0008, Málaga, MA
  - Local Institution - 0002, El Palmar, MU
  - Local Institution - 0003, Valencia, V
  - Local Institution - 0009, A Coruña
  - Local Institution - 0023, Barcelona
  - Local Institution - 0010, Majadahonda

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com